CLINICAL TRIAL: NCT06481709
Title: A Pilot, Phase 1, Randomized, Open-Label, Single-Dose, Four-Way Crossover Study to Compare the Pharmacokinetics of Sapropterin Dihydrochloride 100 mg/mL Oral Suspension (Product Code: RLF-OD032) (Test) With Kuvan® (Sapropterin Dihydrochloride) 100 mg Powder for Oral Solution (Reference) and to Evaluate the Effect of Food and the Effect of Water on the Bioavailability of Sapropterin Dihydrochloride 100 mg/mL Oral Suspension in Healthy Subjects
Brief Title: Study on Sapropterin Dihydrochloride Oral Suspension in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-5439
Record Dates: First submitted 2024-06-06; First posted 2024-07-01 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2023-11

CONDITIONS: Bioavailability
MeSH Terms: interventions — sapropterin

STUDY DESIGN:
Intervention Model Description: In each period, subjects will receive one of the following treatments, according to the randomization scheme:
  Treatment A: 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  Treatment B: 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  Treatment C: 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  Treatment D: 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sequence DCAB (Other): Where the Subject receives in this order
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  Interventions: Drug: RLF-OD032; Drug: Kuvan
- Sequence ADBC (Other): Where the Subject receives in this order
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  Interventions: Drug: RLF-OD032; Drug: Kuvan
- Sequence BACD (Other): Where the Subject receives in this order
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  Interventions: Drug: RLF-OD032; Drug: Kuvan
- Sequence CBDA (Other): Where the Subject receives in this order
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  Interventions: Drug: RLF-OD032; Drug: Kuvan

INTERVENTIONS:
Drug: RLF-OD032 — 100 mg/mL oral suspension
  Other Names: Sapropterin dihydrochloride
Drug: Kuvan — 100 mg powder for oral solution
  Other Names: Sapropterin dihydrochloride

SUMMARY:
This is a single center, Phase 1, randomized, open-label, single-dose, 4 treatment, 4-period, 4-sequence, crossover study designed to compare the pharmacokinetics (PK) of sapropterin from the Test and Reference products, and to evaluate the effect of food and the effect of water administration on the bioavailability of sapropterin from the Test product in healthy subjects.

.

DETAILED DESCRIPTION:
In each period, subjects will receive a single 10 mg/kg dose of sapropterin dihydrochloride on Day 1, under fasting or fed conditions, and with or without water, followed by 24 hours of PK sampling. The study will include a screening visit from Day -30 to Day -1. In each period, eligible subjects will be admitted to the clinical site on Day -1 and will be confined until completion of the assessments on Day 2. There will be a washout period of at least 7 days between doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, light smoker (no more than 10 cigarettes daily) or non smoker, ≥18 and ≤50 years of age, with body mass index (BMI) ≥18.5 and ≤30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 30 days prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Female subjects of non-childbearing potential must be:

   1. post-menopausal (no menstrual period at least 12 consecutive months without any other medical cause and FSH and LH values consistent with being menopausal); or
   2. surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy or tubal ligation) at least 3 months prior to dosing.
4. Sexually active female subjects of childbearing potential must be willing to use an acceptable contraceptive method throughout the study as detailed in the protocol.
5. Willing to take off dentures or mouth piercing at the time of dosing.
6. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Clinically significant abnormal laboratory test results (may be repeated up to two times) or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV)-1 and HIV-2 antibodies at screening.
3. Positive pregnancy test or lactating female subject.
4. Positive urine drug screen.
5. Known allergic reactions to sapropterin dihydrochloride or other related drugs, or to any excipient in the formulation.
6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic blood pressure lower than 90 or over 150 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 bpm) at screening. ECG and vitals signs may be repeated up to two times, to determine if the values are significantly abnormal.
7. Recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
8. History of alcohol addiction requiring treatment.
9. History of abuse of medicinal product or drugs within the last 3 years.
10. History or presence of alcoholism within the last 3 years. (>40 g ethanol/day or more than 10 units per week [1 unit =150 mL of wine, or 360 mL of beer, or 45 mL of 45% alcohol]).
11. Use of medications within the timeframes specified in the protocol
12. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
13. Known predisposition to seizures.
14. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
15. Presence of orthodontic braces or orthodontic retention wires, or any physical findings in the mouth or tongue that would be likely to interfere with successful completion of the dosing procedure.
16. Females who:

    1. Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to study treatment administration.
    2. Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to study treatment administration.
17. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma Medica Research Inc. 4770 Sheppard Ave E,, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence DCAB: The Subject receives in this order
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  RLF-OD032: 100 mg/mL oral suspension
  Kuvan: 100 mg powder for oral solution
- Sequence ADBC: The Subject receives in this order
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  RLF-OD032: 100 mg/mL oral suspension
  Kuvan: 100 mg powder for oral solution
- Sequence BACD: The Subject receives in this order
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  RLF-OD032: 100 mg/mL oral suspension
  Kuvan: 100 mg powder for oral solution
- Sequence CBDA: The Subject receives in this order
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  RLF-OD032: 100 mg/mL oral suspension
  Kuvan: 100 mg powder for oral solution
Period: Overall Study
Arm/Group | Sequence DCAB | Sequence ADBC | Sequence BACD | Sequence CBDA
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 2 | 4
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients Included in the 4 Sequences (DCAB;ADBC;BACD;CBDA): Where the Subject receives these treatments according to the order of the assigned sequence
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  RLF-OD032: 100 mg/mL oral suspension
  Kuvan: 100 mg powder for oral solution
Arm/Group | All Patients Included in the 4 Sequences (DCAB;ADBC;BACD;CBDA)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 16
weight [Mean (Standard Deviation); unit: kg] | 70.4 (10.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25 (4)

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Sapropterin AUC0-t
Description: Area under the concentration-time curve from time zero until the last observed concentration, as calculated by the linear up/log down variant of the trapezoidal method
Time Frame: Time points 1, 0.5, pre-dose (0-hour), and 0.333, 0.667, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16, and 24 hours post-dose.
Population: 2 Subjects didn't complete the treatment phase with C and D
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Treatment A: Where
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
- Treatment B: Where
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
- Treatment C: Where
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
- Treatment D: Where
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 16 | 14 | 14
hr*ng/mL | 989.77 (548.82) | 837.20 (258.17) | 835.52 (276.42) | 791.64 (180.57)

2. Primary Outcome: Baseline-corrected Sapropterin AUC0-t
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 2 Subjects didn't complete the treatment phase with C and D
Measure: Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 16 | 14 | 14
hr*ng/mL | 933.65 (539.81) | 783.15 (251.59) | 780.09 (255.94) | 737.30 (166.92)

3. Primary Outcome: Uncorrected Sapropterin Cmax
Description: Maximum observed concentration
Time Frame: as for outcome 1
Population: 2 Subjects didn't complete the treatment phase with C and D
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 16 | 14 | 14
ng/mL | 170.45 (119.43) | 127.64 (63.98) | 121.92 (60.07) | 127.99 (37.39)

4. Primary Outcome: Baseline-corrected Sapropterin Cmax
Description: Maximum observed concentration
Time Frame: as for outcome 1
Population: 2 Subjects didn't complete the treatment phase with C and D
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 16 | 14 | 14
ng/mL | 168.30 (119.22) | 125.55 (63.74) | 119.81 (59.30) | 125.87 (36.82)

5. Primary Outcome: Uncorrected Sapropterin AUC0-inf
Description: Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: as for outcome 1
Population: 2 Subjects didn't complete the treatment phase with C and D; 1 Subject under treatment B and C not considered due to a concentration-time profiles with the terminal linear phase not clearly defined
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 15 | 13 | 14
hr*ng/mL | 1018.13 (544.08) | 885.12 (257.50) | 848.05 (288.09) | 818.89 (185.13)

6. Primary Outcome: Baseline-corrected Sapropterin AUC0-inf
Description: Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 16 | 15 | 13 | 14
hr*ng/mL | 943.10 (537.40) | 813.04 (254.02) | 783.20 (263.36) | 747.35 (167.02)

ADVERSE EVENTS:
Time Frame: Approximately 30 days (From ICF signature to the last scheduled study procedure)
Groups:
- Treatment A: The Subject receives, according to the assigned sequence, this treatment:
  A is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fasting conditions.
  *RLF-OD032: 100 mg/mL oral suspension
- Treatment B: The Subject receives, according to the assigned sequence, this treatment:
  B is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered without water under fed conditions.
  *RLF-OD032: 100 mg/mL oral suspension
- Treatment C: The Subject receives, according to the assigned sequence, this treatment:
  C is 1 x 10 mg/kg dose* of sapropterin dihydrochloride oral suspension 100 mg/mL administered with water under fed conditions.
  *RLF-OD032: 100 mg/mL oral suspension
- Treatment D: The Subject receives, according to the assigned sequence, this treatment:
  D is 1 x 10 mg/kg dose* of Kuvan (sapropterin dihydrochloride) 100 mg powder for oral solution dissolved in water and administered under fed conditions
  *Kuvan: 100 mg powder for oral solution
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 2/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=16) | Treatment B (N=16) | Treatment C (N=14) | Treatment D (N=14)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT06481709/Prot_SAP_000.pdf